CLINICAL TRIAL: NCT01240031
Title: Framework for Developing Appetising, Energy- and Protein-rich Foods for Patients at Nutritional Risk: Effect on Physiological Functions and Quality of Life
Brief Title: Effect of Energy- and Protein-rich Foods on Physiological Functions and Quality of Life in Undernourished Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Arla Foods (Industry); The Danish Dairy Research Foundation, Denmark (Other)
Responsible Party: Janice Marie Sorensen, Department of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: JMS-2010-29293/19069
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Malnutrition
Keywords: Malnutrition; Nutritional Risk; Intake; Food sensory; Nutritional therapy; Energy; Protein; Handgrip strength; Reaction time; Quality of Life
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Other: Individualised nutritional therapy — Nutritional therapy as based on previous results of the project on patient meal experiences and preferences (note citations below) and comprising of:
  * Thorough sensory and nutrition assessment (questionnaire).
  * Nutrition plan adjusted daily according to the assessment.
  * Serving appetising, energy- and protein-dense meals, snacks and drinks.
Other: Usual nutrition care — Nutritional therapy according to current practice and general nutrition advice.

SUMMARY:
The purpose of this study is to determine whether individualised nutritional therapy comprised of appetising, energy- and protein-rich foods can have a positive effect on physiological function and quality of life of undernourished patients as compared to usual nutrition care.

DETAILED DESCRIPTION:
Undernutrition and insufficent dietary intake in hospitalised patients is a widespread problem. It is associated with increased morbidity and mortality, worsened physiological function and quality of life and increased expenses for the health care system. Food quality has been shown to be positively associated with dietary intake in patients. However, there has lacked knowledge on how food quality can be optimised to promote intake. A project was therefore initiated, which aimed at establishing a framework for developing appetising, energy- and protein-rich foods for patients at nutritional risk. This project included qualitative and quantitative investigation of nutritional risk patients' meal experiences and preferences (se citations below). These results have served as a basis for optimsing energy- and protein-rich foods as part of an indivudalised nutritional therapy aimed at improving dietary intake in nutritional risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Nutritional risk as per Nutrition Risk Screening 2002 (NRS-2002)
* Hospital admited at Rigshospitalets (various medical departments)
* Expect length of stay >= 5 days
* Informed consent to participate

Exclusion Criteria:

* Dementia or other psychiatric condition resulting in an inability to give informed consent and to understand study materials.
* Inability to fairly perform the functional measurements (i.e., handgrip strength, reaction time) due to a hand, wrist, arm, shoulder injury or condition.
* Enteral or parenteral nutrition as primary nutritional therapy.
* Previous participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Intake | Study period during admission in hopsital
  Expressed as energy and protein balance (percent of calculated requirements met by intake as per daily dietary recording)

SECONDARY OUTCOMES:
Handgrip strength | Study period during admission in hopsital
  Grip track dynamometer (3 trials)
Reaction time | Study period during admission in hopsital
  Test for Attentional Performance (TAP version 2, Psytest) Go/NoGo
Quality of life | 28 days
  Short Form 36v2 Health Survey (SF36)

CONTACTS AND LOCATIONS:
Overall Officials: Janice M Sorensen, MSc, Principal Investigator — University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Sorensen JM et al. P155 Food sensory issues in nutritional risk patients: an observational, interview-based study. Clin Nutr Suppl 2009;4(2):91.
- [Background] Sorensen JM et al. OP004 Food sensory issues in nutritional risk patients: a questionnaire study. Clin Nutr Suppl 2010;5(2):2.